CLINICAL TRIAL: NCT03864835
Title: NASH-FITTER: Nonalcoholic Steatohepatitis Fitness Intervention Treatment Targeting Endothelial Dysfunction Reversal
Acronym: NASH-FITTER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Stine, Center Assistant Professor of Medicine and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00012210
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis; NASH - Nonalcoholic Steatohepatitis
Keywords: fatty liver; NASH; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderate intensity aerobic exercise (Experimental): All subjects will undergo DXA and CRF measurement (relative VO2max) under the supervision of an American College of Sports Medicine (ACSM)-certified fitness professional and study physician at the Penn State PM&R Research Laboratories. Subjects selected for the interventional pilot trial will receive a FitBit Charge2 HR and be instructed on how to use a FitBit Hear Rate monitor, Fitbit application, Fitbit website, and Fitabase (secure data management platform utilized by >400 clinical trials). Participants will record their daily food and beverage intake through the Fitbit app. Individualized feedback will be provided by a registered dietician (RD). Subjects that meet requirements for the exercise arm (12 total) will be required to exercise 30 minutes, five days per week at a moderate intensity (HR target corresponding to 45-55% of their relative VO2max). Each session will be supervised in-person at the Penn State University Fitness Center with an ACSM certified exercise physiologist.
  Interventions: Behavioral: Moderate intensity aerobic exercise

INTERVENTIONS:
Behavioral: Moderate intensity aerobic exercise — Subjects that meet requirements for the exercise arm (12 total) will be required to exercise 30 minutes, five days per week at a moderate intensity (HR target corresponding to 45-55% of their relative VO2max). Each session will be supervised in-person at the Penn State University Fitness Center with an ACSM certified exercise physiologist. This is feasible as Zhang et al.(87) found 66 out of 70 subjects (95%) completed the twelve-month supervised in-person moderate-intensity exercise protocol five-days a week.

SUMMARY:
This research is being done to find out if aerobic exercise is beneficial in reversing scarring. Physical activity has been shown to increase fitness in healthy individuals as well as in those with NASH. This research will allow for better understanding the effects of physical activity on fitness and endothelial function in patients with NASH with the goal of reversing scarring.

Approximately 12 people will take part in this research study at Penn State (PSU) Milton S. Hershey Medical Center (HMC), Penn State Physical Medicine & Research (PM&R) Laboratories housed at the Hershey Center for Applied Research (HCAR) and the Penn State University Fitness Center (UFC).

DETAILED DESCRIPTION:
Preliminary studies show universally low cardiorespiratory fitness (CRF) in Nonalcoholic steatohepatitis (NASH) patients was dependent on body composition. The proposed work is based on the hypothesis that gains in cardiorespiratory fitness and improved endothelial function achieved through exercise can arrest or reverse progression of hepatic fibrosis, lessen cardiovascular disease risk (CVD), and improve all-cause mortality in patients with NASH. The aims of this research proposal are designed to characterize and better understand the effects of physical activity (PA) on CRF and endothelial function in patients with NASH. The goal is to arrest progression of fibrosis and reduce CVD risk. This proposal includes a cross-sectional study and a small pilot clinical trial in a high-risk subgroup of NASH most likely to benefit from PA.

ELIGIBILITY:
Inclusion Criteria

•Enrollment and completion of IRB study # 00011797

Exclusion Criteria

* Inability to provide informed consent
* Institutionalized/prisoner
* Non-English-speaking patients due to unavailability of translators for all visits/sessions

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
hepatic fibrosis stage using METAVIR score | 12 months
  The primary endpoint of this study is change in hepatic fibrosis stage.

SECONDARY OUTCOMES:
fibrosis change and gains in cardiorespiratory fitness | 12 months
  correlation between fibrosis change and gains in CRF
flow mediated dilation | 12 months
  correlation between fibrosis change and improvements in FMD
NAFLD Activity Score (NAS) | 12 months
  The diagnosis of nonalcoholic steatohepatitis (NASH) is defined by the presence and pattern of specific histological abnormalities on liver biopsy. A separate system of scoring the features of nonalcoholic fatty liver disease (NA) called the NAFLD Activity Score (NAS) was developed as a tool to measure changes in NAFLD. The grading or NAFLD activity score (NAS) encompasses steatosis, lobular inflammation and ballooning.
intra-hepatic fat content | 12 months
  changes in intra-hepatic fat content
health related quality of life (HRQOL) | 12 months
  PROMIS is a computer adaptive test (CATs) used to assess health related quality of life. The survey contains profiles that measure multiple concepts through a fixed collection of short forms.
Body composition | 12 months
  body composition change

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan G Stine, MD, Principal Investigator — Milton S. Hershey Medical Center

IPD SHARING:
Plan to Share IPD: No